CLINICAL TRIAL: NCT04552964
Title: Assessment of the Impact of an add-on and Its Smartphone Application on the Daily Management of Glaucoma
Acronym: CONDORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CONDORE
Record Dates: First submitted 2020-08-03; First posted 2020-09-17 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: This will be a single centre, single-arm, prospective pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): This will be a single centre, single-arm, prospective pilot study.
  Interventions: Other: Single arm

INTERVENTIONS:
Other: Single arm — Far Best Corrected Visual Acuity (BCVA) ; Intra-Ocular Pressure (IOP) assessment ; Fundus examination ; Automated visual field ; Slit lamp examination ; Pregnancy test ; Patient Satisfaction Questionnaire

SUMMARY:
Glaucoma is one of the most common chronic pathologies and affects several millions patients. Among these, many have a poorly controlled glaucoma, damaging vision and leading to blindness.

One between principal reasons for poor glaucoma medication adherence is forgetfulness. To improve this issue, digital tools may benefit both ophthalmologists and patients by monitoring eye drop administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patient > 18 years old, both genders
2. Diagnosed with glaucoma, with controlled IOP (<18mmHg)
3. Currently receiving a topical glaucoma treatment
4. Receiving a multitherapy a fixed combination of dorzolamide-timolol, preservative-free.
5. Patient willing to participate in the study.
6. Patient familiar with a smartphone and its applications

Exclusion Criteria:

1. Patient with any eye condition in addition to glaucoma requiring expected additional treatment
2. Patient with an ongoing or known history of ocular allergy and/or uveitis and/or viral infection and or ocular infection.
3. Patient who underwent intraocular surgery within the past 3 months or scheduled to undergo intraocular surgery within the next 3 months
4. Patient with best-correct visual acuity <20/70 in the better seeing eye
5. Patient whose drop administration is performed by someone else
6. Alcohol addiction and/or heavy smoker, according to the investigator's judgement.
7. Patient inability to understand the study procedures or to give informed consent.
8. Non-compliant patient (e.g., not willing to attend a visit; way of life interfering with compliance).
9. Participation in this study at the same time as in another clinical study.
10. Patient being institutionalized because of legal or regulatory order, inmate of psychiatric wards, prison or state institutions, or employee of the study sites or of the sponsor's company.
11. Patient not covered by the government health care scheme of the country in which he/she is living (if applicable).
12. Women of childbearing potential, pregnant or breastfeeding: Childbearing potential is defined as a woman who is not using a reliable method of contraception (oral contraceptive, intrauterine device, subcutaneous contraceptive implant, vaginal ring, patch) or is not surgically sterilized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Global patient satisfaction | Week 9
  Global patient satisfaction (Patient satisfaction questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste DERIOT, Dr., Principal Investigator — Centre d'Ophtalmologie Blatin; Emmanuelle ALBERTINI, Dr., Principal Investigator — Centre d'Ophtalmologie Blatin
Locations (1):
- Centre d'Ophtalmologie Blatin, Clermont-Ferrand, France

REFERENCES:
- [Derived] Deriot JB, Albertini E. Is CONNECTDROP(R), a Medication Event Monitoring System Add-On Paired with a Smartphone Application, Acceptable to Patients with Glaucoma for Taking Their Daily Medication? The CONDORE Pilot Study. Ophthalmol Sci. 2024 Apr 30;4(6):100541. doi: 10.1016/j.xops.2024.100541. eCollection 2024 Nov-Dec. PMID 39310045